CLINICAL TRIAL: NCT06538103
Title: Combining Early Lower Eyelid Surgery With Neuromuscular Retraining for Synkinesis Prevention After Facial Palsy.
Brief Title: Eye Soft Surgery for Facial Sinkynesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Arianna Di Stadio, Associate Professor (temporary), University of Catania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UniCT2022
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Facial Paralysis; Sinkynesis
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Kabat therapy home NMR, and eyelid surgery at 90 days (if lagophthalmos with epiphora or ectropion was present)
  Interventions: Procedure: Eye soft surgery; Other: Physical Rehabilitation
- Control (Active Comparator): Kabat therapy and neuromuscular reeducation (NMR) at home
  Interventions: Other: Physical Rehabilitation

INTERVENTIONS:
Procedure: Eye soft surgery — Early lower eyelid surgery will be performed in accordance with the protocol previously described by Di Stadio, with medial or lateral eyelid lifting surgery as indicated. The indication for eye surgery are in case of ectropion (exposure of the conjunctiva due to a reduction in tension of the anterior compartment of the eye muscle) and lagophthalmos (incomplete /abnormal closure of the eye with eyelid in closed position) a lateral lower eyelid lifting surgery is performed. otherwise, in presence of epiphora (the eversion of the lachrymal point) and lagophthalmos medial lower eyelid lifting surgery is done.
  Other Names: Lower eyelid surgery
  Arms: Treatment
Other: Physical Rehabilitation — Kabat therapy and neuromuscular reeducation (NMR) at home Kabat therapy involved thrice-weekly 35-minute sessions.
  Other Names: Kabat

SUMMARY:
Facial synkinesis (FS) is a distressing sequela of facial palsy (FP) characterized by involuntary, simultaneous movements of facial muscles occurring during voluntary facial expressions. Treatment of synkinesis is challenging, and preventive methods are needed.

This study evaluates the efficacy of physical facial nerve rehabilitation (PFNR) therapy alone versus PNFR with eyelid surgery to correct lagophthalmos and prevent the onset of synkinesis.

25 outpatients are randomized to receive either PFNR alone (neuromuscular retraining and Kabat proprioceptive neuromuscular facilitation) or PNFR and early (90 days after FP onset) eyelid surgery (involving a conservative oculoplastic correction for lagophthalmos with epiphora or ectropion). Comprehensive otolaryngological assessments and Magnetic Resonance Imaging (MRI) will be conducted. Synkinesis progression was measured using Another Disease Scale (ADS) at baseline, 3 months 6 months, 12 months, and 24-months post-treatment. The data were analyzed with ANOVA, t-test, Chi-Square analyses.

ELIGIBILITY:
Inclusion Criteria:

* people over 18 years old
* willingness to participate
* acute/new onset of FP (less than 15 days)

Exclusion Criteria:

* neuro-inflammatory diseases (e.g., Multiple Sclerosis)
* FP from systemic disorders (e.g., Guillain-Barré syndrome, Lyme disease, encephalitis)
* FP from middle ear infections or untreated cholesteatoma
* severe cognitive or psychological disorders
* non-consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Sinkinesis | 3, 6, 12, 24 months
  Presence or absence

SECONDARY OUTCOMES:
Recovery of Facial motility | 3, 6, 12, 24 months
  ADS will be used to evaluate the recovery of facial motility
Time to recover facial motility | 3, 6, 12, 24 months
  Evaluation of months needed to recover

CONTACTS AND LOCATIONS:
Overall Officials: Arianna Di Stadio, MD, PhD, Principal Investigator — UniCT
Locations (1):
- Arianna Di Stadio, Catania, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No
The data will be shared after data publication

REFERENCES:
- [Result] Di Stadio A. Eyelid lifting for ectropion and scleral show in facial palsy disease. ORL J Otorhinolaryngol Relat Spec. 2014;76(6):329-35. doi: 10.1159/000369623. Epub 2015 Jan 8. PMID 25572490
- [Result] Di Stadio A. Another Scale for the Assessment of Facial Paralysis? ADS Scale: Our Proposition, How to Use It. J Clin Diagn Res. 2015 Dec;9(12):MC08-11. doi: 10.7860/JCDR/2015/15366.6953. Epub 2015 Dec 1. PMID 26814596
- [Result] Di Stadio A, Gambacorta V, Ralli M, Pagliari J, Longari F, Greco A, Ricci G. Facial taping as biofeedback to improve the outcomes of physical rehab in Bell's palsy: preliminary results of a randomized case-control study. Eur Arch Otorhinolaryngol. 2021 May;278(5):1693-1698. doi: 10.1007/s00405-020-06193-3. Epub 2020 Jul 17. PMID 32681234
- [Result] Monini S, Iacolucci CM, Di Traglia M, Lazzarino AI, Barbara M. Role of Kabat rehabilitation in facial nerve palsy: a randomised study on severe cases of Bell's palsy. Acta Otorhinolaryngol Ital. 2016 Aug;36(4):282-288. doi: 10.14639/0392-100X-783. PMID 27734980
- [Result] Barbara M, Antonini G, Vestri A, Volpini L, Monini S. Role of Kabat physical rehabilitation in Bell's palsy: a randomized trial. Acta Otolaryngol. 2010;130(1):167-72. doi: 10.3109/00016480902882469. PMID 19430987
- [Derived] Di Stadio A, Ralli M, De Luca P, Sossamon J, Frohman TC, Altieri M, La Mantia I, Ferlito S, Frohman EM, Brenner MJ. Combining early lower eyelid surgery with neuromuscular retraining for synkinesis prevention after facial palsy: the role of the eye in aberrant facial nerve regeneration. Front Neurol. 2024 Sep 18;15:1443591. doi: 10.3389/fneur.2024.1443591. eCollection 2024. PMID 39359872